CLINICAL TRIAL: NCT04805333
Title: A Phase 1 Dose Escalation of ArtemiCoffee in Patients With Advanced Ovarian Cancer
Brief Title: Phase 1 Dose Escalation of ArtemiCoffee
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Frederick R. Ueland, M.D. (Other)
Collaborators: ArtemiLife (Unknown)
Responsible Party: Sponsor-Investigator, Frederick R. Ueland, M.D., Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20-GYN-08
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Ovarian Cancer
Keywords: dose escalation; ArtemiCoffee; Artemisia annua; ART-Coffee; herbal
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Dose 1 - 450mg Artemisia annua (Experimental): Participants in this group will consume 1 cup of decaffeinated coffee (450 mg Artemisia annua).
  Interventions: Drug: Artemisia annua 450mg
- Dose 2 - 900mg Artemisia annua (Experimental): Participants in this group will consume 2 cups of decaffeinated coffee (900 mg Artemisia annua).
  Interventions: Drug: Artemisia annua 900mg
- Dose 3 - 1350mg Artemisia annua (Experimental): Participants in this group will consume 3 cups of decaffeinated coffee (1350 mg Artemisia annua).
  Interventions: Drug: Artemisia annua 1350mg
- Dose 5 - 1800mg Artemisia annua (Experimental): Participants in this group will consume 4 cups of decaffeinated coffee (1800 mg Artemisia annua).
  Interventions: Drug: Artemisia annua 1800mg
- Dose Expansion - Recommended Phase II Dose (Experimental): This cohort will be an expansion of 6 patients for further tolerability and secondary endpoints analysis. They will consume the recommended phase II dose (dependent on prior analysis).
  Interventions: Drug: Artemisia annua - recommended phase II dose

INTERVENTIONS:
Drug: Artemisia annua 450mg — Artemisia annua will be self-administered via a preparation of decaffeinated coffee.
  Arms: Dose 1 - 450mg Artemisia annua
Drug: Artemisia annua 900mg — Artemisia annua will be self-administered via a preparation of decaffeinated coffee.
  Arms: Dose 2 - 900mg Artemisia annua
Drug: Artemisia annua 1350mg — Artemisia annua will be self-administered via a preparation of decaffeinated coffee.
  Arms: Dose 3 - 1350mg Artemisia annua
Drug: Artemisia annua 1800mg — Artemisia annua will be self-administered via a preparation of decaffeinated coffee.
  Arms: Dose 5 - 1800mg Artemisia annua
Drug: Artemisia annua - recommended phase II dose — Artemisia annua will be self-administered via a preparation of decaffeinated coffee. The dose for this cohort will be based on analysis of previous cohorts.
  Arms: Dose Expansion - Recommended Phase II Dose

SUMMARY:
This is a phase I dose-escalation study of Artemisia annua (Aa) in patients with advanced ovarian cancer who have completed front-line chemotherapy with carboplatin and paclitaxel. The primary objective of this study is to determine the recommended phase II dose (RP2D) of Artemisia annua.

DETAILED DESCRIPTION:
This is a phase I dose-escalation study of Artemisia annua (Aa) decaffeinated coffee in patients with advanced ovarian cancer who have completed front-line chemotherapy with carboplatin and paclitaxel. The primary objective of this study is to determine the recommended phase II dose (RP2D) of Aa decaf coffee pods. Sequential cohorts of three patients per cohort will have escalating doses of Aa, starting with one cup per day (450mg) and with a maximum of 4 cups per day (1800mg). After identifying the RP2D, the study will evaluate an expansion cohort of 6 patients for further tolerability and secondary endpoints. The secondary endpoints include: 1) Efficacy as measured by time to tumor progression or recurrence; 2) the ability of Aa decaf coffee to influence downstream biomarkers of the NRF2/KEAP1 signaling pathway; and 3) plasma concentrations of artemisinin and dihydroartemisinin.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and willing to sign a written informed consent document.
* Age ≥ 18 years.
* Patients diagnosed with Stage II-IV ovarian cancer who have completed initial first-line therapy with carboplatin and paclitaxel and achieved a complete response.
* Creatinine clearance ≥ 60 mL/min
* Total bilirubin ≤ 1.5 x ULN, and AST and ALT ≤ 3.0 x ULN
* GOG Performance Status ≤ 2.

Exclusion Criteria:

* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study visits, in the opinion of the treating physician.
* Pregnant women are excluded from this study.
* Concurrent use of strong inducers of CYP2A6, including phenobarbital and rifampin
* Women with active gastric ulcers are excluded from this study.
* Patients who are receiving concurrent maintenance therapy with a PARP inhibitor for a known hereditary recombinant deficiency (HRD) mutation. Bevacizumab maintenance therapy is allowed.
* Concurrent use of nevirapine, ritonavir and strong UGT inhibitors or inducers.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2025-02-04 (Actual); Study Completion 2025-02-04 (Actual)

PRIMARY OUTCOMES:
Recommended Phase II Dose | 150 days
  This study will determine the recommended phase II dose of Artemisia annua decaffeinated coffee. Once the dose escalation is finished or 12 patients are evaluated for the dose-limiting toxicity (DLT), the final recommended phase II dose will be determined by isotonic regression to pool the DLT information across all dose levels.

SECONDARY OUTCOMES:
Progression Free Survival | 150 days
  Median progression free survival will be calculated for all groups.

OTHER OUTCOMES:
Change in plasma concentration of artemisinin. | Up to 150 days (baseline and post-treatment)
  The change in plasma concentration of artemisinin will be measured pre- and post-study.
Change in plasma concentration of dihydroartemisinin. | Up to 150 days (baseline and post-treatment)
  The change in plasma concentration of dihydroartemisinin will be measured pre- and post-study.
Change in NQ01 expression. | Up to 150 days (baseline and post-treatment)
  Change in cell-free (cfRNA) levels of NQ01 (NAD(P)H:quinone oxidoreductase 1) will be measured at baseline and post-treatment.
Change in HO-1 expression. | Up to 150 days (baseline and post-treatment)
  Change in cell-free (cfRNA) levels of HO1 (heme oxygenase 1) will be measured at baseline and post-treatment.
Change in ABCF2 expression. | Up to 150 days (baseline and post-treatment)
  Change in cell-free (cfRNA) levels of HO1 (ATP-binding cassette sub-family F member 2) will be measured at baseline and post-treatment.
Change in CD99 expression. | Up to 150 days (baseline and post-treatment)
  Change in cell-free (cfRNA) levels of CD99 (ATP-binding cassette sub-family F member 2) will be measured at baseline and post-treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Ueland, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No